CLINICAL TRIAL: NCT03222505
Title: Development of Walk Assist Device to Improve Community Ambulation
Brief Title: Walk Assist Device to Improve Community Ambulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NUSTU00022438
Record Dates: First submitted 2017-06-22; First posted 2017-07-19 (Actual); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Stroke
Keywords: Stroke; Gait Stride Management Assist; Stroke, post 1 year or longer
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treadmill (Experimental)
  Interventions: Device: Honda Stride Assist Device ON; Other: No Device Worn
- Overground Walking (Experimental)
  Interventions: Device: Honda Stride Assist Device ON; Other: No Device Worn

INTERVENTIONS:
Device: Honda Stride Assist Device ON — Subjects performed assessments of walking and motor performance while wearing the Honda Stride Assist Device.
Other: No Device Worn — Subjects performed assessments of walking and motor performance without wearing the Honda Assist Device.

SUMMARY:
The goal of this research study was to examine the immediate effects of a prototype wearable robotic stride management assist device (SMA) designed by Honda R&D® on clinical walking performance, walking energetics, gait kinematics and corticospinal excitability in individuals with stroke.

DETAILED DESCRIPTION:
The goal of this research study was to examine the immediate effectiveness of a prototype wearable robotic stride management assist device (SMA) designed by Honda R&D on clinical walking performance, walking energetics, gait kinematics and corticospinal excitability in individuals with stroke.

The SMA assists walking by providing a flexion and extension torque assist at the hip joint. The subjects in this study are asked to perform two sets of experiments: one set with the device on and one set with the device turned off. The order in which the subjects performed these sets of experiments is selected randomly. Each set of experiments includes over-ground walking speed and endurance tests, a graded treadmill test with metabolic measures, motion capture and force treadmill analysis, and measures of corticospinal drive using transcranial magnetic stimulation (TMS). The primary outcome to be measured is change in self-selected walking speed with the device on, the secondary outcome measures include metabolic, corticospinal and biomechanical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Stroke subjects with a history of unilateral, supratentorial, ischemic or hemorrhage stroke will be recruited, with lesion location confirmed by radiographic findings.
2. All subjects who score > 10 on the Lower Extremity Motor Score (LEMS) developed previously to measure strength in Spinal Cord Injury (SCI). For the LEMS criteria, preliminary data indicate that subjects with LEMS < 10 in the chronic stages do not recover walking.
3. All subjects will be required to walk > 10 m over ground without physical assistance at self-selected walking speeds ≤ 0.8 m/s using assistive devices and bracing below the knee as needed. A criterion of 0.8 m/s is utilized to target participants with limited or minimal ambulation in the community. Subjects will be further stratified into those who walk < 0.4 m/s and > 0.4 m/s, identified as household vs. limited community ambulators, respectively.
4. Range of motion (ankle: -10 to 30 deg, knee: 0 to 90 deg, hip: -10 to 40 deg) consistent with gait;
5. Medically stable with medical clearance to participate (absence of concurrent illness, including unhealed decubiti, infection, cardiopulmonary disease, osteoporosis, active heterotrophic ossification or peripheral nerve damage in the lower limbs, history of traumatic head injury);
6. Able to tolerate 30 minutes of upright (standing) position without orthostasis (decrease in blood pressure by 20 mmHg systolic and 10 mmHg diastolic; minimized with ambulatory population);
7. Must not be undergoing concurrent physical therapy to eliminate effects of additional interventions;
8. Patients prescribed medications for spasticity will not be excluded from participation but will be asked to maintain current levels of medication or inform the researcher if changes are necessary.

   -

Exclusion Criteria:

1. Women of childbearing potential will not be excluded, although women who are pregnant will be excluded due to potential forces at trunk from body weight support or pelvic assistance;
2. Significant cardiorespiratory or metabolic disease that may limit exercise participation.
3. Weights limit > 250 lbs (limit of most counter-weight safety systems).
4. History of previous orthopedic or neurological conditions which may impair walking.
5. Exclusion for TMS: pacemaker, metal implants in the head region, history of epilepsy or seizures, skull fractures or skull deficits, concussion within the last 6 months, unexplained recurring headaches, medications that lower seizure threshold, and pregnancy.
6. Subjects with scores < 23 on the Mini Mental Status Exam will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-01; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Start With Device ON: Participants in this arm first completed testing with the device on, then repeated the testing a week later with the device turned off.
- Start With Device OFF: Participants in this arm first completed testing with the device off, then repeated the testing a week later with the device turned on.
Period: Overall Study
Arm/Group | Start With Device ON | Start With Device OFF
Started | 5 | 7
Completed | 5 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Start With Device ON | Start With Device OFF | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (8.2) | 59.9 (6.3) | 57.8 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 4 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 12
Self-Selected Walking Speed less than 0.8 m/s [Mean (Standard Deviation); unit: meters per second] — Participants needed to have a self-selected walking speed of 0.8 m/s or less for a distance of ten meters or greater.
  meters per second | 0.57 (0.21) | 0.62 (0.17) | 0.60 (0.18)

OUTCOME MEASURES:

1. Primary Outcome: Change in Six Minute Walk Test Between Device Turned ON and OFF - Distance Traveled
Description: The 6 Minute Walk Test (6MWT) is a test of endurance, by measuring the distance a subject can walk indoors on a flat, hard surface in a period of 6 minutes, using assistive devices, as necessary.The distance is measured with a measuring wheel. The instructions are "Walk covering as much ground as you can in 6 min. You can stop to sit or stand if needed."
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: feet
Groups:
- Device ON: Data collected from while the device was turned on.
- Device OFF: Data collected from while the device was turned off.
Arm/Group | Device ON | Device OFF
Number analyzed (Participants) | 12 | 12
feet | 837.1 (342.2) | 804.8 (358.5)

2. Primary Outcome: Change in Peak Treadmill (TM) Velocity Between Device Turned ON and OFF - Self Selected Walking Speed
Description: Peak treadmill (TM) velocity: subjects walked on motorized treadmill with harness but no Body Weight Support (BWS). Testing started at 0.5 km/h and was increased in 0.5 km/h increments every 3 minutes until peak TM speed was achieved (identified as ability to sustain speed for ≥1min without stopping the treadmill).
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Device ON | Device OFF
Number analyzed (Participants) | 12 | 12
meters per second | 0.95 (0.28) | 0.84 (0.30)

3. Secondary Outcome: Percent Change in Excitability of Transcranial Magnetic Stimulation (TMS) Rectus Femoris (RF) Between Device ON and Device OFF
Description: TMS measurements will involve generating motor evoked potentials (MEP) for each muscle from two different coil positions - 2cm on either side of the vertex. Motor evoked potentials (MEPs) at intensities ranging from 70 - 140% active threshold will be generated for each muscle from each coil position. TMS is a safe, non-invasive, painless method of brain stimulation that has been widely used to study the physiology of the representations of muscles in the motor cortex in healthy and neurologically disordered individuals. A positive percent change in excitability indicates higher excitability in the device-on condition. A negative percent change in excitability indicates higher excitability in the device-off condition.
Time Frame: Day 1
Population: Device ON and Device OFF arms were combined as the interest of this metric was the change in excitability between device on and device off conditions within a participant.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Difference Between Device ON and Device OFF: Difference in excitability for device on and off.
Arm/Group | Difference Between Device ON and Device OFF
Number analyzed (Participants) | 12
percent change | 19.02 (34.5)

4. Secondary Outcome: Change in Percent Excitability of Transcranial Magnetic Stimulation (TMS), Dorsiflexor Tibialis Anterior (TA) Between Device ON and Device OFF
Description: as for outcome 3
Time Frame: Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Difference Between Device ON and Device OFF
Number analyzed (Participants) | 12
percent change | -13.53 (31.6)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assessed, before and after every data collection session, through study completion, an average of 2 days.
Groups:
- Device ON: The arm reflects time during study participation when the participants were wearing the device.
- Device OFF: The arm reflects time during study participation when the participants were not wearing the device.
Arm/Group | Device ON | Device OFF
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-04-16): https://cdn.clinicaltrials.gov/large-docs/05/NCT03222505/Prot_SAP_000.pdf